CLINICAL TRIAL: NCT01675544
Title: PRospective Evaluation of Electrocardiographic Voltage Changes and Six Minute Walk Test for Predicting Readmissions in Heart Failure (PREEMT-HF Study)
Acronym: PREEMT-HF
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Other Study IDs: 12-16350
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Heart Failure
Keywords: Heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure Admission: Patients admitted for acute decompensated heart failure
  Interventions: Procedure: Electrocardiogram; Procedure: Six minute walk test

INTERVENTIONS:
Procedure: Electrocardiogram — EKG voltage changes between admission and discharge
  Other Names: EKG
Procedure: Six minute walk test
  Other Names: 6-MWT

SUMMARY:
Purpose of the study: To identify whether Electrocardiographic QRS voltage changes (between admission and pre-discharge) and pre discharge 6- minute walk test in patients admitted with acute heart failure can identify patients at risk for recurrent admissions for heart failure.

DETAILED DESCRIPTION:
Primary Objective Determine the ability of EKG voltage changes and pre discharge 6-minute walk test (6-MWT) to predict repeat heart failure hospitalization (HFH) in patients admitted with acute decompensated heart failure (ADHF).

Secondary Objectives

1. Determine the ability of EKG voltage changes and pre discharge 6-MWT) to predict a composite of 1 year mortality and HFH in patients admitted with ADHF.
2. Determine the ability of proportionate pulse pressure, orthostatic blood pressure changes and pre discharge inferior vena cava (IVC) diameter by portable ultrasound to predict HFH and mortality

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age, admitted with a diagnosis of ADHF and fulfilling the following criteria:

  1. Evidence of systemic congestion (manifested by any 2 of the following criteria: jugular venous distension, edema, pulmonary rales, Left ventricular S3, or radiographic evidence of pulmonary venous congestion)
  2. Elevated Brain natriuretic peptide
  3. Need for at least 1 dose of intravenous loop diuretic

Exclusion Criteria:

* Cardiogenic shock, Acute coronary syndromes (patients with mild elevation in troponin related to heart failure will not be excluded), patients who are admitted for another principal problem and develop ADHF in the hospital, pregnant females, end stage renal disease on hemodialysis, expected survival < 6 months.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with acute decompensated heart failure
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Venkata M Alla, MBBS, Principal Investigator — Creighton University
Locations (1):
- Creighton University Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Heart Failure Admission: Patients admitted for acute decompensated heart failure
  Electrocardiogram: EKG voltage changes between admission and discharge
  Six minute walk test
Period: Overall Study
Arm/Group | Heart Failure Admission
Started | 46
Completed | 44
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Heart Failure Admission
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Emergency Room Visit or Hospitalization for Acute Decompensated Heart Failure (ADHF)
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Heart Failure Admission
Number analyzed (Participants) | 44
participants | 20

2. Primary Outcome: Mortality
Description: All cause mortality at 1 year
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Heart Failure Admission
Number analyzed (Participants) | 44
participants | 9

ADVERSE EVENTS:
Arm/Group | Heart Failure Admission
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes